CLINICAL TRIAL: NCT04089709
Title: Well-arm Exercise in Distal Radius Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Trent Guthrie, Principal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11912
Record Dates: First submitted 2019-09-12; First posted 2019-09-13 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Distal Radius Fracture
Keywords: Distal radius fracture; cross-education; immobilization
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups, treatment or no treatment. Randomizations will be balanced at random accrual points.
Who Masked: Outcomes Assessor
Masking Description: Patients will be randomized using an online randomization tool. Study folders will be placed in order and include the consent form and exercise sheet if randomized to the treatment group. Those randomized to the control group will be given an information sheet on distal radius fractures. Patients will be consented by an unblinded research assistant in order for the treating physician to remain blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study arm (Experimental): Patients randomized to this group will be provided exercises to perform with the uninjured arm once daily for 3 months.
  Interventions: Behavioral: Well-arm Exercise
- Control arm (No Intervention): Patients randomized to this group will not be provided exercises for the "well-arm" and will be managed according to the current standard of care.

INTERVENTIONS:
Behavioral: Well-arm Exercise — Patients randomized to the treatment arm will perform these exercises on the contralateral arm once daily for 3 months: wrist flexion and extension, ball or sock squeeze, wrist curls and biceps curls. Participants allocated to this study arm will be provided a print out of the exercises with detailed explanations and pictures of each exercise.
  Arms: Study arm

SUMMARY:
A single center randomized control study. Patients >18 years with isolated distal radius fractures treated non-operatively will be randomly assigned to either the treatment group (exercise of contralateral "well" arm) or control group (standard fracture care and rehabilitation).

DETAILED DESCRIPTION:
Distal radius fractures are common injuries, especially in the aging population. Fracture healing requires immobilization of the injury, which inevitably leads to muscle atrophy and joint stiffness. This strength lost during immobilization can be problematic in patients who are already de-conditioned at baseline. Previous research using healthy participants found that exercising a non-immobilized, "well", arm helped attenuate muscle atrophy in the contralateral immobilized arm. The study aims to answer the following questions: Does exercise of the contralateral arm prevent muscle atrophy and weakness of the injured arm? Does exercise of the contralateral arm improve pain scores in the injured arm

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years with an isolated distal radius fracture treated non-operatively

Exclusion Criteria:

* Operative treatment, additional injures, previous injury to same arm, neuropathy or neuromuscular disease, dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-11-30 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Grip strength | 3 months
  Grip strength will be measured using a dynamometer at all clinic visits.
Forearm Circumference | 3 months
  Forearm circumference will be measured at the widest point of the forearm, approximately 2cm distal to the elbow. This measurement will be taken at all clinic visits.

SECONDARY OUTCOMES:
Pain scores of injured arm. | 3 months
  A visual analog scale (VAS) score will be collected at the first and all subsequent clinic visits.

OTHER OUTCOMES:
Wrist Range of Motion | 3 months
  Range of motion of the injured wrist will be measured after the period of immobilization.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart T Guthrie, MD, Principal Investigator — Henry Ford Hospital System
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States